CLINICAL TRIAL: NCT03261336
Title: A Phase II Study of Oral Calcitriol in Combination With Ketoconazole in Castration Resistant Prostate Cancer, Progressing Despite Primary ADT and Abiraterone
Brief Title: Oral Calcitriol With Ketoconazole in CRPC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: can not meet enrollment
Sponsor: Donald Trump, MD (Other)
Responsible Party: Sponsor-Investigator, Donald Trump, MD, CEO & Executive Director, Inova Schar Cancer Institute, Inova Health Care Services
Organization: Inova Health Care Services (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-2200
Record Dates: First submitted 2017-07-12; First posted 2017-08-25 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Castration-resistant Prostate Cancer
MeSH Terms: interventions — Calcitriol; Ketoconazole; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Calcitriol 10mcg QD X3, weekly + Ketoconazole 400mg po TID and Hydrocortisone 20mg AM, 10mg PM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Calcitriol, Ketoconazole, Hydrocortisone (Experimental): Patients receive calcitriol (10mcg QD X3 weekly) in addition to ketoconazole (400mg QD) and hydrocortisone (20mg AM, 10 mg PM).
  Interventions: Drug: Calcitriol, Ketoconazole, Hydrocortisone

INTERVENTIONS:
Drug: Calcitriol, Ketoconazole, Hydrocortisone — Calcitriol (0.5 mcg caplets) given in escalating doses, orally QD X3 consecutive days every week Ketoconazole, 200 mg tablets, 2 tablets orally TID Hydrocortisone 20mg AM, 10mg PM orally starting in the evening before the first dose of Calcitriol
  Other Names: Rocaltrol®; active form of vitamin D3

SUMMARY:
The aim of this study is to estimate the PSA response rate with the use of ketoconazole (400mg QD + hydrocortisone 20mg AM, 10 mg PM) among men with CRPC in whom disease has progressed despite abiraterone

DETAILED DESCRIPTION:
This study will aim to describe objective tumor responses to the combination of oral calcitriol and ketoconazole and hydrocortisone-among patients with measurable disease using modified RECIST 1.1 criteria.

Additionally, we will determine toxicities, and tolerability of oral calcitriol combination with daily oral ketoconazole, and hydrocortisone in this patient population.

this is a single arm phase II trial of ketoconazole (400mg QD + hydrocortisone 20mg AM, 10 mg PM) among men with CRPC in whom disease has progressed despite abiraterone

ELIGIBILITY:
Inclusion Criteria

For inclusion in the trial, a patient must fulfill all of the following criteria:

1. Greater than or equal to 18 years of age. The effects of ketoconazole and high-dose calcitriol have not been studied adequately in patients <18 years of age and prostate cancer has not been described in children.
2. Histologically or cytologically confirmed adenocarcinoma consistent clinically with androgen Independent prostate cancer
3. Measurable disease with elevated PSA or evaluable disease (PSA elevation will constitute evaluable disease).
4. No cytotoxic chemotherapy for extensive disease prior to study entry will be allowed; given the recent data regarding the role of docetaxel + ADT in patients beginning ADT for advanced disease, such "adjuvant chemotherapy will be allowed (no more than 6 cycles) retinoids, vitamin D analogues, PPAR agonists or antagonists, antiandrogens, progestational agents, estrogens, PC-SPES, LHRH analogues, vaccines, cytokines will not be considered "cytotoxics." Patients who have previously received ketoconazole + glucocorticoids will NOT be eligible for this trial.
5. Patients who have received antiandrogens or progestational agents as therapy for prostate cancer must discontinue therapy and demonstrate a rising PSA > 28 days following discontinuation (antiandrogen withdrawal - AAW) (>42 days for bicalutamide or nilutamide). Patients who receive megestrol acetate as therapy for "hot flashes" at a dose of <40mg per day may continue this therapy during this trial. The dose of the megestrol acetate should not be changed during protocol treatment. Patients undergoing androgen deprivation using LHRH analogues must continue such agents or undergo orchiectomy to maintain castrate levels of testosterone.
6. Patients must have prostate cancer that is advanced or recurrent.
7. Patients should not have received any chemotherapy or investigational agents for at least 28 days before entering the study.
8. Eastern Clinical Oncology Group performance status 0 or 1
9. Life expectancy >3 months.
10. Patients must have normal organ and marrow function as defined below:

    leukocytes: >3,000/μl hemoglobin: > 8 g/dl absolute neutrophil count (ANC):>1,500/μl platelets: >75,000/μl total bilirubin: within normal institutional limit AST/ALT: <2.5 X institutional upper limit of normal creatinine: < 2mg/dL calcium: not above normal institutional limit
11. Patients should be able to receive oral medications.
12. Patients with brain metastases which are stable and have been treated with surgery and/or irradiation will be eligible for this trial.
13. The effects of high-dose calcitriol and ketoconazole on the developing human fetus are unknown. For this reason and because these agents as well are known to be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform the treating physician immediately.
14. Ability to understand and the willingness to sign a written informed consent document.
15. Progressive disease must have occurred on abiraterone within the prior 12 months and patient must not have received treatment with enzalutamide.

Men of all ethnic groups are eligible for this trial. Efforts will be made to include minority groups and all representative ethnicities and races in the community.

Exclusion Criteria

Any of the following is a criterion for exclusion from the trial:

1. Known severe hypersensitivity to ketoconazole, calcitriol or any of the excipients of these products.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to calcitriol, ketoconazole, or other agents used in study.
3. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial.
4. History of kidney, ureteral, or bladder stones within the last 5 years
5. Heart failure or significant heart disease including significant arrhythmias, myocardial infarction within the last 3 months, unstable angina, documented ejection fraction <30%, or current digoxin therapy.
6. Thiazide therapy within 7 days from entering the study.
7. Requirement for concurrent systemic glucocorticoid therapy at greater than physiologic replacement doses
8. Unwillingness to stop calcium supplementation.
9. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) or intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Human immunodeficiency virus-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible PK interactions with ketoconazole or other agents administered during the study. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
11. Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St John's wort, alfentanil, alfuzosin, almotriptan, alprazolam, amiodarone, amitriptyline, amprenavir, aprepitant, aripiprazole, bepridil, bortezomib, bosentan, budesonide, buprenorphine, buspirone, carbamazepine, cilostazol, cisapride, cyclosporine, delavirdine, didanosine, digoxin, disopyramidedofetilide, donepezil, eletriptan, eplerenone, fluticasone, fosamprenavir, galantamine, systemic griseofulvin, indinavir, levobupivacaine, lopinavir, midazolam, mifepristone, modafinil, nateglinide, nefazadone, nelfinavir, oxcarbazepine, pimozide, quetiapine, quinidine, repaglinide, rifabutin, rifampin, rifapentine, ritonavir, saquinavir, sildenafil, sirolimus, tacrolimus, tadalafil, tolterodine, theophyllines, tolterodine, triazolam, valdecoxib, vardenafil, ziprasidone, zonisamide, statins, with the exception of pravastatin (Pravachol) or other "statins" which are not metabolized by or induce CYP3A4, calcium channel blockers, and macrolides or other agents that will be significantly perturbed in a clinically important way by the P450 inhibitory properties of ketoconazole
12. Concomitant use of proton pump inhibitors or H2 blockers
13. Treatment with a non-approved or investigational drug or agent within 28 days before day 1 of trial treatment.
14. Any unresolved chronic toxicity greater then CTC Grade 2 from previous anticancer therapy.
15. Incomplete healing from previous oncologic treatments or other major surgery.
16. Inability to swallow oral capsules.
17. Patients on digoxin will be excluded from this study.

Products Dosage and Mode of Administration

* Ketoconazole, 200 mg tablets, 2 tablets orally TID
* Calcitriol (0.5 mcg caplets) given in escalating doses, orally QD X3 consecutive days every week
* Hydrocortisone 20mg AM, 10mg PM orally starting in the evening before the first dose of Calcitriol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Skip (Donald) Trump, MD, Principal Investigator — CEO & Executive Director Inova Schar Cancer Institute
Locations (1):
- Inova Schar Cancer Institute, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bikle DD, Pillai S. Vitamin D, calcium, and epidermal differentiation. Endocr Rev. 1993 Feb;14(1):3-19. doi: 10.1210/edrv-14-1-3. No abstract available. PMID 8491153
- [Background] McElwain MC, Dettlebach MA, Modzelewski RA, et al. Antiproliferative effects in vitro and in vivo of 1,25-dihydroxyvitamin D3 and a vitamin D3 analog in a squamous cell carcinoma model system Mol Cell Diff 3 (1) 31 (1995).
- [Background] Modzelewski RA. Apoptotic effects of paclitaxel and calcitriol in rat dunning MLL and human PC-3 prostate tumor cells in vitro. Proc Amer Assoc Cancer Res 40 580, 1999.
- [Background] Hershberger PA, Yu WD, Modzelewski RA, Rueger RM, Johnson CS, Trump DL. Calcitriol (1,25-dihydroxycholecalciferol) enhances paclitaxel antitumor activity in vitro and in vivo and accelerates paclitaxel-induced apoptosis. Clin Cancer Res. 2001 Apr;7(4):1043-51. PMID 11309356
- [Background] Light BW, Yu WD, McElwain MC, Russell DM, Trump DL, Johnson CS. Potentiation of cisplatin antitumor activity using a vitamin D analogue in a murine squamous cell carcinoma model system. Cancer Res. 1997 Sep 1;57(17):3759-64. PMID 9288784
- [Background] Hershberger PA, Modzelewski RA, Shurin ZR, Rueger RM, Trump DL, Johnson CS. 1,25-Dihydroxycholecalciferol (1,25-D3) inhibits the growth of squamous cell carcinoma and down-modulates p21(Waf1/Cip1) in vitro and in vivo. Cancer Res. 1999 Jun 1;59(11):2644-9. PMID 10363987
- [Background] McGuire TF, Trump DL, Johnson CS. Vitamin D(3)-induced apoptosis of murine squamous cell carcinoma cells. Selective induction of caspase-dependent MEK cleavage and up-regulation of MEKK-1. J Biol Chem. 2001 Jul 13;276(28):26365-73. doi: 10.1074/jbc.M010101200. Epub 2001 Apr 30. PMID 11331275
- [Background] McGuire TF, Trump DL and Johnson CS. 1,25-dihydroxyvitamin D3 induces cytosolic accumulation of MEKK-1 before onset of apoptosis in a p38 MAPK-regulated manner. Proc. Amer. Assoc. Cancer Res. 2159, 435 (2002).
- [Background] Hershberger PA, McGuire TF, Yu WD, Zuhowski EG, Schellens JH, Egorin MJ, Trump DL, Johnson CS. Cisplatin potentiates 1,25-dihydroxyvitamin D3-induced apoptosis in association with increased mitogen-activated protein kinase kinase kinase 1 (MEKK-1) expression. Mol Cancer Ther. 2002 Aug;1(10):821-9. PMID 12492115
- [Background] Johnson CS, Egorin MJ, Zuhowski R, 35 al. Effects of high dose calcitriol (1,25 dihydroxyvitamin D3) on the pharmacokinetics of paclitaxel or carboplatin: results of two phase I studies Amer Soc Clin Oncol 19 210a (2000).
- [Background] Muindi JR, Peng Y, Potter DM, Hershberger PA, Tauch JS, Capozzoli MJ, Egorin MJ, Johnson CS, Trump DL. Pharmacokinetics of high-dose oral calcitriol: results from a phase 1 trial of calcitriol and paclitaxel. Clin Pharmacol Ther. 2002 Dec;72(6):648-59. doi: 10.1067/mcp.2002.129305. PMID 12496746
- [Background] Muindi JR, Modzelewski RA, Peng Y, Hershberger PA, Trump DL and Johnson CS. Plasma 1, 25-dihydroxycholecalciferol pharmacokinetics in normal and tumor bearing mice. Oncology (in press).
- [Background] Yu WD, McElwain MC, Modzelewski RA, Russell DM, Smith DC, Trump DL, Johnson CS. Enhancement of 1,25-dihydroxyvitamin D3-mediated antitumor activity with dexamethasone. J Natl Cancer Inst. 1998 Jan 21;90(2):134-41. doi: 10.1093/jnci/90.2.134. PMID 9450573
- [Background] Bernardi RJ, Trump DL, Yu WD, McGuire TF, Hershberger PA, Johnson CS. Combination of 1alpha,25-dihydroxyvitamin D(3) with dexamethasone enhances cell cycle arrest and apoptosis: role of nuclear receptor cross-talk and Erk/Akt signaling. Clin Cancer Res. 2001 Dec;7(12):4164-73. PMID 11751517
- [Background] Klein RG, Arnaud SB, Gallagher JC, Deluca HF, Riggs BL. Intestinal calcium absorption in exogenous hypercortisonism. Role of 25-hydroxyvitamin D and corticosteroid dose. J Clin Invest. 1977 Jul;60(1):253-9. doi: 10.1172/JCI108762. PMID 874087
- [Background] Ahmed S, Johnson CS, Rueger RM, Trump DL. Calcitriol (1,25-dihydroxycholecalciferol) potentiates activity of mitoxantrone/dexamethasone in an androgen independent prostate cancer model. J Urol. 2002 Aug;168(2):756-61. PMID 12131364
- [Background] Hershberger PA, Modzelewski RA, Rueger RM, Blum KE, Trump DL, and Johnson CS. Enhanced anti-tumor efficacy with dexamethasone/calcitriol/cisplatin therapy: role of P21WAF1. Proc. Amer. Assoc. Cancer Res. 41, 15 (2000).
- [Background] Yu WD, Rueger RM, Fuller RW, Johnson CS, and Trump DL. 1,25-dihydroxycholecalciferol (calcitriol) enhancement of chemotherapeutic efficacy: synergistic effects by median dose effect. Proc. Amer. Assoc. Cancer Res. 42, 84 (2001).
- [Background] Trump DL, Serafine S, Brufsky J, et al. High dose calcitriol (1,25(OH)2 vitamin D3) + dexamethasone in androgen independent prostate cancer (AIPC). Amer Soc Clin Oncol 19 337a (2000).
- [Background] Omdahl JL, Bobrovnikova EA, Choe S, Dwivedi PP, May BK. Overview of regulatory cytochrome P450 enzymes of the vitamin D pathway. Steroids. 2001 Mar-May;66(3-5):381-9. doi: 10.1016/s0039-128x(00)00157-4. PMID 11179747
- [Background] Feldman D. Ketoconazole and other imidazole derivatives as inhibitors of steroidogenesis. Endocr Rev. 1986 Nov;7(4):409-20. doi: 10.1210/edrv-7-4-409. No abstract available. PMID 3536461
- [Background] Reinhardt TA, Horst RL. Ketoconazole inhibits self-induced metabolism of 1,25-dihydroxyvitamin D3 and amplifies 1,25-dihydroxyvitamin D3 receptor up-regulation in rat osteosarcoma cells. Arch Biochem Biophys. 1989 Aug 1;272(2):459-65. doi: 10.1016/0003-9861(89)90240-3. PMID 2546501
- [Background] Evans RM. The steroid and thyroid hormone receptor superfamily. Science. 1988 May 13;240(4854):889-95. doi: 10.1126/science.3283939.
- [Background] Darwish HM, DeLuca HF. Recent advances in the molecular biology of vitamin D action. Prog Nucleic Acid Res Mol Biol. 1996;53:321-44. doi: 10.1016/s0079-6603(08)60149-x. PMID 8650307
- [Background] Christakos S, Raval-Pandya M, Wernyj RP, Yang W. Genomic mechanisms involved in the pleiotropic actions of 1,25-dihydroxyvitamin D3. Biochem J. 1996 Jun 1;316 ( Pt 2)(Pt 2):361-71. doi: 10.1042/bj3160361. PMID 8687373
- [Background] Darwish H, DeLuca HF. Vitamin D-regulated gene expression. Crit Rev Eukaryot Gene Expr. 1993;3(2):89-116. PMID 8391882
- [Background] Studzinski GP, McLane JA, Uskokovic MR. Signaling pathways for vitamin D-induced differentiation: implications for therapy of proliferative and neoplastic diseases. Crit Rev Eukaryot Gene Expr. 1993;3(4):279-312. PMID 8286848
- [Background] Weigel NL. Steroid hormone receptors and their regulation by phosphorylation. Biochem J. 1996 Nov 1;319 ( Pt 3)(Pt 3):657-67. doi: 10.1042/bj3190657. PMID 8920964
- [Background] Norman AW, Nemere I, Zhou LX, Bishop JE, Lowe KE, Maiyar AC, Collins ED, Taoka T, Sergeev I, Farach-Carson MC. 1,25(OH)2-vitamin D3, a steroid hormone that produces biologic effects via both genomic and nongenomic pathways. J Steroid Biochem Mol Biol. 1992 Mar;41(3-8):231-40. doi: 10.1016/0960-0760(92)90349-n. PMID 1314073
- [Background] Slater SJ, Kelly MB, Taddeo FJ, Larkin JD, Yeager MD, McLane JA, Ho C, Stubbs CD. Direct activation of protein kinase C by 1 alpha,25-dihydroxyvitamin D3. J Biol Chem. 1995 Mar 24;270(12):6639-43. doi: 10.1074/jbc.270.12.6639. PMID 7896803
- [Background] de Boland AR, Morelli S, Boland R. 1,25(OH)2-vitamin D3 signal transduction in chick myoblasts involves phosphatidylcholine hydrolysis. J Biol Chem. 1994 Mar 25;269(12):8675-9. PMID 8132595
- [Background] Khare S, Tien XY, Wilson D, Wali RK, Bissonnette BM, Scaglione-Sewell B, Sitrin MD, Brasitus TA. The role of protein kinase-C alpha in the activation of particulate guanylate cyclase by 1 alpha,25-dihydroxyvitamin D3 in CaCo-2 cells. Endocrinology. 1994 Jul;135(1):277-83. doi: 10.1210/endo.135.1.7912183.
- [Background] de Boland AR, Norman A. Evidence for involvement of protein kinase C and cyclic adenosine 3',5' monophosphate-dependent protein kinase in the 1,25-dihydroxy-vitamin D3-mediated rapid stimulation of intestinal calcium transport, (transcaltachia). Endocrinology. 1990 Jul;127(1):39-45. doi: 10.1210/endo-127-1-39. PMID 2163320
- [Background] Gniadecki R. Activation of Raf-mitogen-activated protein kinase signaling pathway by 1,25-dihydroxyvitamin D3 in normal human keratinocytes. J Invest Dermatol. 1996 Jun;106(6):1212-7. doi: 10.1111/1523-1747.ep12348498. PMID 8752659
- [Background] MacDonald PN, Baudino TA, Tokumaru H, Dowd DR, Zhang C. Vitamin D receptor and nuclear receptor coactivators: crucial interactions in vitamin D-mediated transcription. Steroids. 2001 Mar-May;66(3-5):171-6. doi: 10.1016/s0039-128x(00)00200-2. PMID 11179724
- [Background] Barletta F, Freedman LP, Christakos S. Enhancement of VDR-mediated transcription by phosphorylation: correlation with increased interaction between the VDR and DRIP205, a subunit of the VDR-interacting protein coactivator complex. Mol Endocrinol. 2002 Feb;16(2):301-14. doi: 10.1210/mend.16.2.0764. PMID 11818502
- [Background] Zhang C, Dowd DR, Staal A, Gu C, Lian JB, van Wijnen AJ, Stein GS, MacDonald PN. Nuclear coactivator-62 kDa/Ski-interacting protein is a nuclear matrix-associated coactivator that may couple vitamin D receptor-mediated transcription and RNA splicing. J Biol Chem. 2003 Sep 12;278(37):35325-36. doi: 10.1074/jbc.M305191200. Epub 2003 Jul 2. PMID 12840015
- [Background] Herdick M, Carlberg C. Agonist-triggered modulation of the activated and silent state of the vitamin D(3) receptor by interaction with co-repressors and co-activators. J Mol Biol. 2000 Dec 15;304(5):793-801. doi: 10.1006/jmbi.2000.4267. PMID 11124027
- [Background] Colston KW, Chander SK, Mackay AG, Coombes RC. Effects of synthetic vitamin D analogues on breast cancer cell proliferation in vivo and in vitro. Biochem Pharmacol. 1992 Aug 18;44(4):693-702. doi: 10.1016/0006-2952(92)90405-8. PMID 1324683
- [Background] Frappart L, Falette N, Lefebvre MF, Bremond A, Vauzelle JL, Saez S. In vitro study of effects of 1,25 dihydroxyvitamin D3 on the morphology of human breast cancer cell line BT.20. Differentiation. 1989 Mar;40(1):63-9. doi: 10.1111/j.1432-0436.1989.tb00814.x. PMID 2545494
- [Background] Shabahang M, Buras RR, Davoodi F, Schumaker LM, Nauta RJ, Evans SR. 1,25-Dihydroxyvitamin D3 receptor as a marker of human colon carcinoma cell line differentiation and growth inhibition. Cancer Res. 1993 Aug 15;53(16):3712-8. PMID 8393379
- [Background] Mangelsdorf DJ, Koeffler HP, Donaldson CA, Pike JW, Haussler MR. 1,25-Dihydroxyvitamin D3-induced differentiation in a human promyelocytic leukemia cell line (HL-60): receptor-mediated maturation to macrophage-like cells. J Cell Biol. 1984 Feb;98(2):391-8. doi: 10.1083/jcb.98.2.391. PMID 6319426
- [Background] Godyn JJ, Xu H, Zhang F, Kolla S, Studzinski GP. A dual block to cell cycle progression in HL60 cells exposed to analogues of vitamin D3. Cell Prolif. 1994 Jan;27(1):37-46. doi: 10.1111/j.1365-2184.1994.tb01404.x. PMID 10465025
- [Background] Rigby WF, Noelle RJ, Krause K, Fanger MW. The effects of 1,25-dihydroxyvitamin D3 on human T lymphocyte activation and proliferation: a cell cycle analysis. J Immunol. 1985 Oct;135(4):2279-86. PMID 2993410
- [Background] Wang QM, Jones JB, Studzinski GP. Cyclin-dependent kinase inhibitor p27 as a mediator of the G1-S phase block induced by 1,25-dihydroxyvitamin D3 in HL60 cells. Cancer Res. 1996 Jan 15;56(2):264-7. PMID 8542578
- [Background] Liu M, Lee MH, Cohen M, Bommakanti M, Freedman LP. Transcriptional activation of the Cdk inhibitor p21 by vitamin D3 leads to the induced differentiation of the myelomonocytic cell line U937. Genes Dev. 1996 Jan 15;10(2):142-53. doi: 10.1101/gad.10.2.142. PMID 8566748
- [Background] Biggs JR, Kraft AS. Inhibitors of cyclin-dependent kinase and cancer. J Mol Med (Berl). 1995 Oct;73(10):509-14. doi: 10.1007/BF00198902. PMID 8581512
- [Background] Sherr CJ, Roberts JM. Inhibitors of mammalian G1 cyclin-dependent kinases. Genes Dev. 1995 May 15;9(10):1149-63. doi: 10.1101/gad.9.10.1149. No abstract available. PMID 7758941
- [Background] Sheikh MS, Rochefort H, Garcia M. Overexpression of p21WAF1/CIP1 induces growth arrest, giant cell formation and apoptosis in human breast carcinoma cell lines. Oncogene. 1995 Nov 2;11(9):1899-905. PMID 7478620
- [Background] Henkart PA. ICE family proteases: mediators of all apoptotic cell death? Immunity. 1996 Mar;4(3):195-201. doi: 10.1016/s1074-7613(00)80428-8. No abstract available. PMID 8624810
- [Background] Hockenbery DM. The bcl-2 oncogene and apoptosis. Semin Immunol. 1992 Dec;4(6):413-20. PMID 1286168
- [Background] Simboli-Campbell M, Narvaez CJ, Tenniswood M, Welsh J. 1,25-Dihydroxyvitamin D3 induces morphological and biochemical markers of apoptosis in MCF-7 breast cancer cells. J Steroid Biochem Mol Biol. 1996 Jul;58(4):367-76. doi: 10.1016/0960-0760(96)00055-6. PMID 8903420
- [Background] Xu HM, Tepper CG, Jones JB, Fernandez CE, Studzinski GP. 1,25-Dihydroxyvitamin D3 protects HL60 cells against apoptosis but down-regulates the expression of the bcl-2 gene. Exp Cell Res. 1993 Dec;209(2):367-74. doi: 10.1006/excr.1993.1322. PMID 8262155
- [Background] Henry HL. The 25(OH)D(3)/1alpha,25(OH)(2)D(3)-24R-hydroxylase: a catabolic or biosynthetic enzyme? Steroids. 2001 Mar-May;66(3-5):391-8. doi: 10.1016/s0039-128x(00)00158-6. PMID 11179748
- [Background] Miller GJ, Stapleton GE, Hedlund TE, Moffat KA. Vitamin D receptor expression, 24-hydroxylase activity, and inhibition of growth by 1alpha,25-dihydroxyvitamin D3 in seven human prostatic carcinoma cell lines. Clin Cancer Res. 1995 Sep;1(9):997-1003. PMID 9816072
- [Background] Bareis P, Bises G, Bischof MG, Cross HS, Peterlik M. 25-hydroxy-vitamin d metabolism in human colon cancer cells during tumor progression. Biochem Biophys Res Commun. 2001 Jul 27;285(4):1012-7. doi: 10.1006/bbrc.2001.5289. PMID 11467853
- [Background] Zhao J, Tan BK, Marcelis S, Verstuyf A, Bouillon R. Enhancement of antiproliferative activity of 1alpha,25-dihydroxyvitamin D3 (analogs) by cytochrome P450 enzyme inhibitors is compound- and cell-type specific. J Steroid Biochem Mol Biol. 1996 Feb;57(3-4):197-202. doi: 10.1016/0960-0760(95)00256-1. PMID 8645629
- [Background] Peehl DM, Seto E, Hsu JY, Feldman D. Preclinical activity of ketoconazole in combination with calcitriol or the vitamin D analogue EB 1089 in prostate cancer cells. J Urol. 2002 Oct;168(4 Pt 1):1583-8. doi: 10.1097/01.ju.0000030158.18335.84. PMID 12352462
- [Background] Ly LH, Zhao XY, Holloway L, Feldman D. Liarozole acts synergistically with 1alpha,25-dihydroxyvitamin D3 to inhibit growth of DU 145 human prostate cancer cells by blocking 24-hydroxylase activity. Endocrinology. 1999 May;140(5):2071-6. doi: 10.1210/endo.140.5.6698. PMID 10218956
- [Background] Strom M, Sandgren ME, Brown TA, DeLuca HF. 1,25-Dihydroxyvitamin D3 up-regulates the 1,25-dihydroxyvitamin D3 receptor in vivo. Proc Natl Acad Sci U S A. 1989 Dec;86(24):9770-3. doi: 10.1073/pnas.86.24.9770. PMID 2481316
- [Background] Chen TL, Cone CM, Morey-Holton E, Feldman D. Glucocorticoid regulation of 1,25(OH)2-vitamin D3 receptors in cultured mouse bone cells. J Biol Chem. 1982 Nov 25;257(22):13564-9. No abstract available. PMID 6292196
- [Background] Levy J, Zuili I, Yankowitz N, Shany S. Induction of cytosolic receptors for 1 alpha, 25-dihydroxyvitamin D3 in the immature rat uterus by oestradiol. J Endocrinol. 1984 Mar;100(3):265-9. doi: 10.1677/joe.0.1000265. PMID 6321624
- [Background] Petkovich PM, Heersche JN, Tinker DO, Jones G. Retinoic acid stimulates 1,25-dihydroxyvitamin D3 binding in rat osteosarcoma cells. J Biol Chem. 1984 Jul 10;259(13):8274-80. PMID 6330107
- [Background] Reinhardt TA, Horst RL. Parathyroid hormone down-regulates 1,25-dihydroxyvitamin D receptors (VDR) and VDR messenger ribonucleic acid in vitro and blocks homologous up-regulation of VDR in vivo. Endocrinology. 1990 Aug;127(2):942-8. doi: 10.1210/endo-127-2-942. PMID 2164926
- [Background] Bouillon R, Okamura WH, Norman AW. Structure-function relationships in the vitamin D endocrine system. Endocr Rev. 1995 Apr;16(2):200-57. doi: 10.1210/edrv-16-2-200. No abstract available. PMID 7781594
- [Background] Trump DL, Havlin KH, Messing EM, Cummings KB, Lange PH, Jordan VC. High-dose ketoconazole in advanced hormone-refractory prostate cancer: endocrinologic and clinical effects. J Clin Oncol. 1989 Aug;7(8):1093-8. doi: 10.1200/JCO.1989.7.8.1093. PMID 2474059
- [Background] OH WK. Secondary hormonal therapies in the treatment of prostate cancer. Urology. 2002 Sep;60(3 Suppl 1):87-92; discussion 93. doi: 10.1016/s0090-4295(02)01581-9. PMID 12231058
- [Background] Hirst M, Feldman D. Glucocorticoids down-regulate the number of 1, 25-dihydroxyvitamin D3 receptors in mouse intestine. Biochem Biophys Res Commun. 1982 Apr 29;105(4):1590-6. doi: 10.1016/0006-291x(82)90970-6. No abstract available. PMID 6285911
- [Background] Kimberg DV, Baerg RD, Gershon E, Graudusius RT. Effect of cortisone treatment on the active transport of calcium by the small intestine. J Clin Invest. 1971 Jun;50(6):1309-21. doi: 10.1172/JCI106610. PMID 4325312
- [Background] Haynes RC. Agents affecting calcification: calcium, parathyroid hormone, calcitonin, vitamin D, and other compounds. The Pharmacological Basis of Therapeutics. Gilman AG, Rall TW, Nies AS, Taylor P (eds). New York Pergamon Press 1496 (1990).
- [Background] Fakih M, Johnson CS, Trump DL. Glucocorticoids and treatment of prostate cancer: a preclinical and clinical review. Urology. 2002 Oct;60(4):553-61. doi: 10.1016/s0090-4295(02)01741-7. No abstract available. PMID 12385906
- [Background] Nishimura K, Nonomura N, Satoh E, Harada Y, Nakayama M, Tokizane T, Fukui T, Ono Y, Inoue H, Shin M, Tsujimoto Y, Takayama H, Aozasa K, Okuyama A. Potential mechanism for the effects of dexamethasone on growth of androgen-independent prostate cancer. J Natl Cancer Inst. 2001 Nov 21;93(22):1739-46. doi: 10.1093/jnci/93.22.1739. PMID 11717335
- [Background] Tannock IF, Osoba D, Stockler MR, Ernst DS, Neville AJ, Moore MJ, Armitage GR, Wilson JJ, Venner PM, Coppin CM, Murphy KC. Chemotherapy with mitoxantrone plus prednisone or prednisone alone for symptomatic hormone-resistant prostate cancer: a Canadian randomized trial with palliative end points. J Clin Oncol. 1996 Jun;14(6):1756-64. doi: 10.1200/JCO.1996.14.6.1756. PMID 8656243
- [Background] Kantoff PW, Halabi S, Conaway M, Picus J, Kirshner J, Hars V, Trump D, Winer EP, Vogelzang NJ. Hydrocortisone with or without mitoxantrone in men with hormone-refractory prostate cancer: results of the cancer and leukemia group B 9182 study. J Clin Oncol. 1999 Aug;17(8):2506-13. doi: 10.1200/JCO.1999.17.8.2506. PMID 10561316
- [Background] Small EJ, Meyer M, Marshall ME, Reyno LM, Meyers FJ, Natale RB, Lenehan PF, Chen L, Slichenmyer WJ, Eisenberger M. Suramin therapy for patients with symptomatic hormone-refractory prostate cancer: results of a randomized phase III trial comparing suramin plus hydrocortisone to placebo plus hydrocortisone. J Clin Oncol. 2000 Apr;18(7):1440-50. doi: 10.1200/JCO.2000.18.7.1440. PMID 10735891
- [Background] Cunningham D, Gilchrist NL, Cowan RA, Forrest GJ, McArdle CS, Soukop M. Alfacalcidol as a modulator of growth of low grade non-Hodgkin's lymphomas. Br Med J (Clin Res Ed). 1985 Oct 26;291(6503):1153-5. doi: 10.1136/bmj.291.6503.1153. PMID 2996693
- [Background] Koeffler HP, Hirji K, Itri L. 1,25-Dihydroxyvitamin D3: in vivo and in vitro effects on human preleukemic and leukemic cells. Cancer Treat Rep. 1985 Dec;69(12):1399-407. PMID 2416438
- [Background] Rolla D, Paoletti E, Marsano L, Mulas D, Peloso G, Cannella G. Effects of subcutaneous calcitriol administration on plasma calcium and parathyroid hormone concentrations in continuous ambulatory peritoneal dialysis uremic patients. Perit Dial Int. 1993;13(2):118-21. PMID 8494932
- [Background] Davies M. High-dose vitamin D therapy: indications, benefits and hazards. Int J Vitam Nutr Res Suppl. 1989;30:81-6. PMID 2507709
- [Background] Smith DC, Johnson CS, Freeman CC, Muindi J, Wilson JW, Trump DL. A Phase I trial of calcitriol (1,25-dihydroxycholecalciferol) in patients with advanced malignancy. Clin Cancer Res. 1999 Jun;5(6):1339-45. PMID 10389917
- [Background] Beer TM, Munar M, Henner WD. A Phase I trial of pulse calcitriol in patients with refractory malignancies: pulse dosing permits substantial dose escalation. Cancer. 2001 Jun 15;91(12):2431-9. PMID 11413535
- [Background] Beer TM, Eilers KM, Garzotto M, Egorin MJ, Lowe BA, Henner WD. Weekly high-dose calcitriol and docetaxel in metastatic androgen-independent prostate cancer. J Clin Oncol. 2003 Jan 1;21(1):123-8. doi: 10.1200/jco.2003.05.117. PMID 12506180
- [Background] Kaufmann SH, Desnoyers S, Ottaviano Y, Davidson NE, Poirier GG. Specific proteolytic cleavage of poly(ADP-ribose) polymerase: an early marker of chemotherapy-induced apoptosis. Cancer Res. 1993 Sep 1;53(17):3976-85. PMID 8358726
- [Background] Paul A, Wilson S, Belham CM, Robinson CJ, Scott PH, Gould GW, Plevin R. Stress-activated protein kinases: activation, regulation and function. Cell Signal. 1997 Sep;9(6):403-10. doi: 10.1016/s0898-6568(97)00042-9. PMID 9376221
- [Background] Lewis TS, Shapiro PS, Ahn NG. Signal transduction through MAP kinase cascades. Adv Cancer Res. 1998;74:49-139. doi: 10.1016/s0065-230x(08)60765-4. No abstract available. PMID 9561267
- [Background] Levrero M, De Laurenzi V, Costanzo A, Gong J, Wang JY, Melino G. The p53/p63/p73 family of transcription factors: overlapping and distinct functions. J Cell Sci. 2000 May;113 ( Pt 10):1661-70. doi: 10.1242/jcs.113.10.1661. PMID 10769197
- [Background] Yu WD, Chang MJ, Trump DL, Johnson CS. Interleukin-1alpha synergistic in vivo enhancement of cyclophosphamide- and carboplatin-mediated antitumor activity. Cancer Immunol Immunother. 1997 Aug;44(6):316-22. doi: 10.1007/s002620050388. PMID 9298933
- [Background] Kim D, Gregory CW, French FS, Smith GJ, Mohler JL. Androgen receptor expression and cellular proliferation during transition from androgen-dependent to recurrent growth after castration in the CWR22 prostate cancer xenograft. Am J Pathol. 2002 Jan;160(1):219-26. doi: 10.1016/S0002-9440(10)64365-9. PMID 11786415
- [Background] Gregory CW, Kim D, Ye P, D'Ercole AJ, Pretlow TG, Mohler JL, French FS. Androgen receptor up-regulates insulin-like growth factor binding protein-5 (IGFBP-5) expression in a human prostate cancer xenograft. Endocrinology. 1999 May;140(5):2372-81. doi: 10.1210/endo.140.5.6702. PMID 10218991
- [Background] Smitherman AB, Mohler JL, Maygarden SJ, Ornstein DK. Expression of annexin I, II and VII proteins in androgen stimulated and recurrent prostate cancer. J Urol. 2004 Feb;171(2 Pt 1):916-20. doi: 10.1097/01.ju.0000104674.70170.cd. PMID 14713853
- [Background] Smitherman AB, Gregory CW, Mohler JL. Apoptosis levels increase after castration in the CWR22 human prostate cancer xenograft. Prostate. 2003 Sep 15;57(1):24-31. doi: 10.1002/pros.10271. PMID 12886520
- [Background] Mohler JL, Morris TL, Ford OH 3rd, Alvey RF, Sakamoto C, Gregory CW. Identification of differentially expressed genes associated with androgen-independent growth of prostate cancer. Prostate. 2002 Jun 1;51(4):247-55. doi: 10.1002/pros.10086. PMID 11987153
- [Background] Kurahashi I, Matsunuma A, Kawane T, Abe M, Horiuchi N. Dexamethasone enhances vitamin D-24-hydroxylase expression in osteoblastic (UMR-106) and renal (LLC-PK1) cells treated with 1alpha,25-dihydroxyvitamin D3. Endocrine. 2002 Mar;17(2):109-18. doi: 10.1385/ENDO:17:2:109. PMID 12041912
- [Background] Akeno N, Matsunuma A, Maeda T, Kawane T, Horiuchi N. Regulation of vitamin D-1alpha-hydroxylase and -24-hydroxylase expression by dexamethasone in mouse kidney. J Endocrinol. 2000 Mar;164(3):339-48. doi: 10.1677/joe.0.1640339. PMID 10694374
- [Background] Kang S, Li XY, Duell EA, Voorhees JJ. The retinoid X receptor agonist 9-cis-retinoic acid and the 24-hydroxylase inhibitor ketoconazole increase activity of 1,25-dihydroxyvitamin D3 in human skin in vivo. J Invest Dermatol. 1997 Apr;108(4):513-8. doi: 10.1111/1523-1747.ep12289736. PMID 9077483
- [Background] Schuster I, Egger H, Bikle D, Herzig G, Reddy GS, Stuetz A, Stuetz P, Vorisek G. Selective inhibition of vitamin D hydroxylases in human keratinocytes. Steroids. 2001 Mar-May;66(3-5):409-22. doi: 10.1016/s0039-128x(00)00159-8. PMID 11179750
- [Background] Sakaki T, Sawada N, Abe D, Komai K, Shiozawa S, Nonaka Y, Nakagawa K, Okano T, Ohta M, Inouye K. Metabolism of 26,26,26,27,27,27-F6-1alpha,25-dihydroxyvitamin D3 by CYP24: species-based difference between humans and rats. Biochem Pharmacol. 2003 Jun 15;65(12):1957-65. doi: 10.1016/s0006-2952(03)00190-4. PMID 12787875
- [Background] Elbashir SM, Harborth J, Weber K, Tuschl T. Analysis of gene function in somatic mammalian cells using small interfering RNAs. Methods. 2002 Feb;26(2):199-213. doi: 10.1016/S1046-2023(02)00023-3. PMID 12054897
- [Background] Kuo MH, Allis CD. In vivo cross-linking and immunoprecipitation for studying dynamic Protein:DNA associations in a chromatin environment. Methods. 1999 Nov;19(3):425-33. doi: 10.1006/meth.1999.0879. PMID 10579938
- [Background] Smith ML. Mdm2 sensitizes MCF7 breast cancer cells to cisplatin or carboplatin. Breast Cancer Res Treat. 1999 Nov;58(2):99-105. doi: 10.1023/a:1006390107197. PMID 10674873
- [Background] Fillippovich I, Sorokina N, Gatei M, Haupt Y, Hobson K, Moallem E, Spring K, Mould M, McGuckin MA, Lavin MF, Khanna KK. Transactivation-deficient p73alpha (p73Deltaexon2) inhibits apoptosis and competes with p53. Oncogene. 2001 Jan 25;20(4):514-22. doi: 10.1038/sj.onc.1204118. PMID 11313982
- [Background] Mandic A, Viktorsson K, Molin M, Akusjarvi G, Eguchi H, Hayashi SI, Toi M, Hansson J, Linder S, Shoshan MC. Cisplatin induces the proapoptotic conformation of Bak in a deltaMEKK1-dependent manner. Mol Cell Biol. 2001 Jun;21(11):3684-91. doi: 10.1128/MCB.21.11.3684-3691.2001. PMID 11340162
- [Background] Mabuchi S, Ohmichi M, Kimura A, Hisamoto K, Hayakawa J, Nishio Y, Adachi K, Takahashi K, Arimoto-Ishida E, Nakatsuji Y, Tasaka K, Murata Y. Inhibition of phosphorylation of BAD and Raf-1 by Akt sensitizes human ovarian cancer cells to paclitaxel. J Biol Chem. 2002 Sep 6;277(36):33490-500. doi: 10.1074/jbc.M204042200. Epub 2002 Jun 26. PMID 12087097
- [Background] Hisamoto K, Ohmichi M, Kanda Y, Adachi K, Nishio Y, Hayakawa J, Mabuchi S, Takahashi K, Tasaka K, Miyamoto Y, Taniguchi N, Murata Y. Induction of endothelial nitric-oxide synthase phosphorylation by the raloxifene analog LY117018 is differentially mediated by Akt and extracellular signal-regulated protein kinase in vascular endothelial cells. J Biol Chem. 2001 Dec 14;276(50):47642-9. doi: 10.1074/jbc.M103853200. Epub 2001 Oct 10. PMID 11595733
- [Background] Dent P, Grant S. Pharmacologic interruption of the mitogen-activated extracellular-regulated kinase/mitogen-activated protein kinase signal transduction pathway: potential role in promoting cytotoxic drug action. Clin Cancer Res. 2001 Apr;7(4):775-83. No abstract available. PMID 11309321
- [Background] Agoulnik IU, Krause WC, Bingman WE 3rd, Rahman HT, Amrikachi M, Ayala GE, Weigel NL. Repressors of androgen and progesterone receptor action. J Biol Chem. 2003 Aug 15;278(33):31136-48. doi: 10.1074/jbc.M305153200. Epub 2003 May 27. PMID 12771131
- [Background] Cadepond F, Ulmann A, Baulieu EE. RU486 (mifepristone): mechanisms of action and clinical uses. Annu Rev Med. 1997;48:129-56. doi: 10.1146/annurev.med.48.1.129. PMID 9046951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was closed at site in 2018 due to enrollment challenges. Only 1 patient was enrolled to trial. No evaluable results.
Period: Overall Study
Arm/Group | Calcitriol, Ketoconazole, Hydrocortisone
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Calcitriol, Ketoconazole, Hydrocortisone
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 78 [78 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: Assessment of PSA every 4 weeks
Time Frame: 2 years
Population: Only one patient enrolled to study and was discontinued early due to AE.
Arm/Group | Calcitriol, Ketoconazole, Hydrocortisone
Number analyzed (Participants) | 0

2. Secondary Outcome: Tumor Response
Description: Objective tumor response among patients with measurable disease using modified RECIST1.1
Time Frame: 2 years
Population: Only one patient was enrolled and was discontinued due to AE.
Arm/Group | Calcitriol, Ketoconazole, Hydrocortisone
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicity and Tolerability of Experimental Arm
Description: Descriptive analysis of observed toxicity and patient reports of tolerating experimental treatment
Time Frame: 2 years
Population: Patient developed hypercalcemia and was discontinued from study. AE is known, not unexpected.
Measure: Count of Participants; unit: Participants
Arm/Group | Calcitriol, Ketoconazole, Hydrocortisone
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: AE data was collected on a single patient during one month in 2017.
Description: Definition consistent with clinicaltrials.gov
Arm/Group | Calcitriol, Ketoconazole, Hydrocortisone
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol, Ketoconazole, Hydrocortisone (N=1)
hypercalcemia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was closed due to inability to accrue. One patient was entered on study and did develop hypercalcemia which led to treatment discontinuation. Insufficient time on study to evaluate response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT03261336/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT03261336/Prot_SAP_001.pdf